CLINICAL TRIAL: NCT01745224
Title: Revlite Laser System Compared to the Candela Alex TriVantage System Refractory Mixed Type Melasma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped because patient enrollment requirements were not met.
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN12-REV-TRI-AK
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: This was a comparative study where the device was used outside of the recommended treatment usage. It was used to assess the Revlite device for feasibility and not health outcomes.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Revlite Q switched Nd:YAG laser (Experimental): Revlite Q switched Nd:YAG laser 1064 nm
  Interventions: Device: Revlite Q switched Nd:YAG; Device: Trivantage Q switched Nd: YAG
- TriVantage Q switched Nd:YAG laser (Experimental): TriVantage Q switched Nd:YAG laser 1064nm
  Interventions: Device: Revlite Q switched Nd:YAG; Device: Trivantage Q switched Nd: YAG

INTERVENTIONS:
Device: Revlite Q switched Nd:YAG — Revlite Q switched Nd:YAG 1064nm
Device: Trivantage Q switched Nd: YAG — Trivantage Q switched Nd: YAG 1064nm

SUMMARY:
This proof of concept study will be conducted to assess the aesthetic improvement in refractory mixed type melasma in subjects treated with two FDA 510K approved devices: Q Switched Nd: YAG Laser vs. Alex TriVantage

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Fitzpatrick Skin Type III-VI
2. Subjects with mixed (epidermal and dermal) type melasma diagnosed by Wood's Lamp.
3. Subjects who are over the age of 18 years of age
4. The subject is willing and able to comply with study instructions and return to the clinic for required visits.
5. The subject's melasma has persisted for greater than 6 months and has failed to respond to conventional treatment with hydroquinone cream or other topical lightening agents.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject has a history of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis.
3. The subject has any skin pathology or condition that could interfere with the evaluation or requires the use of interfering topical or systemic therapy.
4. The subject has an uncorrected coagulation defect or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 30 days prior to entering this study.
7. The subject has used photosensitizing drugs (e.g., Declomycin, sulfa antibiotics, phenothiazines, etc.) within a timeframe where photosensitization from these drugs may still be present.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has Diabetes Type 1 or 2.
11. The subject has a sensitivity to hydroquinone or Retin-A.
12. The subject has evidence of a compromised immune system or hepatitis.
13. Has had microdermabrasion in past 3 months, other laser or Intense Pulsed Light treatment or chemical peels to the face in past 6 months, injectable fillers, topical retinoids, over-the-counter anti-aging products past 2 weeks.
14. Has a history of keloids or hypertrophic scarring
15. Has permanent make-up and/or is unwilling to refrain from using semi-permanent cosmetics during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Changes in Melasma Determined by Physician | 3 months post last treatment
  The Global Aesthetic Improvement scale was used to determine the amount of improvement. This scale ranges from 1 to 5, where 1 is very much improved, 2 is much improved, 3 is improved, 4 is no change, and 5 is worsened.

SECONDARY OUTCOMES:
Universal Pain Scale for Subject Tolerability | 3 months post last treatment
  The subject pain tolerability was assessed using the Universal Pain Scale. This scale ranges from 0 (no pain) to 10 (worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- NY Laser and Skin Care, New York, New York, United States